CLINICAL TRIAL: NCT04712032
Title: A PHASE III, RANDOMISED CONTROLLED TRIAL ASSESSING THE VALUE OF INDOCYANINE GREEN IN THE LEAKAGE RATE OF COLORECTAL ANASTOMOSES
Brief Title: Anastomotic Leakage and Value Of Indocyanine Green in Decreasing Leakage Rates
Acronym: AVOID
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Catharina Ziekenhuis Eindhoven (Other); Haga Hospital (Other); Jeroen Bosch Ziekenhuis (Other); Amphia Hospital (Other); Alrijne Hospital (Other); IJsselland (Unknown)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P19.079
Record Dates: First submitted 2021-01-14; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Colo-rectal Cancer; Crohn Disease; Resectable Colorectal Carcinoma
MeSH Terms: conditions — Colonic Neoplasms; Crohn Disease

STUDY DESIGN:
Intervention Model Description: National randomized controlled trial.
Who Masked: Participant
Masking Description: Intraoperative imaging is unable to blind the surgeon. Patient is only blinded preoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Image Guided Bowel Anastomosis group (Experimental): ICG-guided perfusion assessment
  Interventions: Drug: ICG-guided bowel perfusion assessment
- Conventional Bowel Anastomosis group (No Intervention): conventional perfusion assessment

INTERVENTIONS:
Drug: ICG-guided bowel perfusion assessment — ICG will be injected prior to anastomosis creation, to assess perfusion status of the bowel.
  Arms: Image Guided Bowel Anastomosis group

SUMMARY:
Anastomotic leakage (AL) is one of the major complications after gastrointestinal surgery. Compromised tissue perfusion at the anastomosis site increases the risk of AL. Indocyanine green (ICG) combined with fluorescent near infrared imaging has proven to be a feasible and reproducible application for real-time intraoperative quantification of the tissue perfusion and cohort studies showed reduced leakage rate. Unfortunately, these studies were not randomized. Therefore, we propose a nationwide randomized controlled trial to identify the value of ICG for AL in colorectal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for laparoscopic or robotic-assisted colorectal resection with primary anastomosis;
2. Patients aged over 18 years old;
3. Has the ability to communicate well with the Investigator in the Dutch language and willing to comply with the study restrictions;
4. Signed informed consent prior to any study-mandated procedure;

Exclusion Criteria:

1. Known allergy or history of adverse reaction to ICG, iodine or iodine dyes;
2. Severe liver or kidney insufficiency;
3. Hyperthyroidism or a benign thyroid tumour;
4. Pregnant or breastfeeding women;
5. Scheduled for palliative surgery or terminal ill
6. Scheduled for a diverting stoma
7. Any condition that the investigator considers to be potentially jeopardizing the patients well-being or the study objectives (following a detailed medical history and physical examination;
8. Subject taking phenobarbital, phenylbutazone, primidone, phenytoin, haloperidol, nitrofurantoin, probenecid;
9. Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 978 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
90-days Anastomotic Leakage (AL) rate | 90 days
  Anastomotic leakage rate

SECONDARY OUTCOMES:
30-days Anastomotic Leakage ( AL) rate | 30 days
  Anastomotic leakage rate
complication rate | 90 days
mortality | 90 days
days in hospital stay | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Vahrmeijer, MD, PhD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faber RA, Meijer RPJ, Droogh DHM, Jongbloed JJ, Bijlstra OD, Boersma F, Braak JPBM, Meershoek-Klein Kranenbarg E, Putter H, Holman FA, Mieog JSD, Neijenhuis PA, van Staveren E, Bloemen JG, Burger JWA, Aukema TS, Brouwers MAM, Marinelli AWKS, Westerterp M, Doornebosch PG, van der Weijde A, Bosscha K, Handgraaf HJM, Consten ECJ, Sikkenk DJ, Burggraaf J, Keereweer S, van der Vorst JR, Hutteman M, Peeters KCMJ, Vahrmeijer AL, Hilling DE. Indocyanine green near-infrared fluorescence bowel perfusion assessment to prevent anastomotic leakage in minimally invasive colorectal surgery (AVOID): a multicentre, randomised, controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2024 Oct;9(10):924-934. doi: 10.1016/S2468-1253(24)00198-5. Epub 2024 Aug 13. PMID 39151436
- [Derived] Meijer RPJ, Faber RA, Bijlstra OD, Braak JPBM, Meershoek-Klein Kranenbarg E, Putter H, Mieog JSD, Burggraaf K, Vahrmeijer AL, Hilling DE; AVOID study group. AVOID; a phase III, randomised controlled trial using indocyanine green for the prevention of anastomotic leakage in colorectal surgery. BMJ Open. 2022 Apr 1;12(4):e051144. doi: 10.1136/bmjopen-2021-051144. PMID 35365509